CLINICAL TRIAL: NCT05310565
Title: The Effects of Chiropractic Care on the Quality of Life and Autonomic Nervous System in Adults With Colon Cancer: a Single-arm Pilot Trial
Brief Title: The Effects of Chiropractic in Adults With Colon Cancer
Acronym: CCX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Life University (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I-0019
Record Dates: First submitted 2022-03-07; First posted 2022-04-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Colon Cancer Stage III; Colon Cancer Stage IV
Keywords: Chiropractic; Colon Cancer; Spinal manipulation; Autonomic nervous system; CEA; patient reported outcomes
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-Arm pilot
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiropractic (Experimental): Cervical chiropractic care
  Interventions: Procedure: HVLA cervical chiropractic adjustments

INTERVENTIONS:
Procedure: HVLA cervical chiropractic adjustments — Chiropractic high velocity low amplitude adjustment

SUMMARY:
The main objectives of this single-arm pilot trial are to investigate the feasibility of our protocol in terms of 1) recruitment, 2) adherence, 3) tolerability, 4) acceptability and 5) retention. We aim to recruit 20 participants with advanced colon cancer (stage 3-4) who will have assessments of their autonomic nervous system function, carcinoembryonic antigen (CEA) levels, and patient-reported outcomes. Thereafter, patients will be directed to a nearby field clinic to receive twice-weekly cervical assessments & high-velocity, low-amplitude (HVLA) cervical adjustments for a period of 6 weeks. Re-assessments will be performed following 2 weeks and 6 weeks of chiropractic care.

DETAILED DESCRIPTION:
After providing informed consent, individuals will undergo 6 weeks of chiropractic care. Throughout these 6 weeks there will be three assessments (Day 1, Week 2, and Week 6) that each include the following:

1. Isometric hand grip
2. Postural challenge
3. Patient-reported outcome surveys
4. Off-site blood draw for CEA level testing (only Day 0 and Week 6)

Each assessment will consist of the following recordings:

1. Electrodermal activity [EDA]
2. Impedance cardiography [ICG]
3. Electrocardiogram [ECG]

ELIGIBILITY:
Inclusion Criteria:

* Males & females 18 years of age or older
* Able to provide informed consent
* Diagnosed with stage 3 or stage 4 colon cancer and currently receiving standard of care with a medical doctor.

Exclusion Criteria:

* Individuals with a known disorder resulting in syncope/fainting during postural changes (e.g., POTS, orthostatic hypotension)
* Cancer has metastasized to the cervical spine
* Individuals who have had a serious injury or surgery to the head, torso, lower body within the past 6 months.
* Individuals with evidence or medical history of clinically significant psychiatric disorder like anti-social disorder, schizophrenia, or borderline personality disorder that is uncontrolled or untreated.
* Individuals who currently have pending health related legal litigation.
* Individuals with a known heart condition (e.g., arrhythmia) that could result in an aberrant electrocardiogram.
* Individuals with a pacemaker
* Individuals who are on short benzodiazepines which include midazolam & triazolam
* Individuals with conditions that could result in neck instability such as rheumatoid arthritis.
* Individuals who do not present with a subluxation in the upper cervical region (C1/C2) at any point during the 6 weeks of chiropractic care.
* Individuals with a condition that may cause weak or brittle bones such as osteoporosis
* Since x-rays may be requested for care, participants who are pregnant will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Upon reaching target number of completed participant trials
  Length of time needed to recruit target number of participants
Patient adherence rate | Upon reaching target number of completed participant trials
  Proportion of participants able to adhere to the testing & treatment protocol/schedule
Patient tolerability rate | Upon reaching target number of completed participant trials
  Proportion of participants able to perform all aspects of the testing regimen
Acceptability of treatment regimen to participants | Week 6
  8-item Theoretical Framework of Acceptability questionnaire
Patient Retention | Upon reaching target number of completed participant trials
  Proportion of enrolled participants who complete the full trial

SECONDARY OUTCOMES:
Electrodermal activity (EDA) skin conductance level (SCL) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) skin conductance level (SCL) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) skin conductance level (SCL) | Week 6
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Week 6
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 6
  2 sensors on first and second digits of non-dominant hand
Impedance cardiogram (ICG) pre-ejection period (PEP) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 6
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 6
  2 sensors on chest and 2 sensors on back
ECG interbeat interval | Day 1
  3 sensors on torso
ECG interbeat interval | Week 2
  3 sensors on torso
ECG interbeat interval | Week 6
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Day 1
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 2
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 6
  3 sensors on torso
ECG de-trended fluctuation analysis | Day 1
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 2
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 6
  3 sensors on torso
Carcinoembryonic antigen (CEA) levels | Day 1
  Off-site blood draw and lab testing
Carcinoembryonic antigen (CEA) levels | Week 6
  Off-site blood draw and lab testing
Patient-reported outcomes | Day 0
  5 questionnaires: EORTC QLQ-C30, COMPASS-31, PROMIS-29, PROMIS-Cog, Perceived Stress Scale
Patient-reported outcomes | Day 1
  5 questionnaires: EORTC QLQ-C30, COMPASS-31, PROMIS-29, PROMIS-Cog, Perceived Stress Scale
Patient-reported outcomes | Week 2
  5 questionnaires: EORTC QLQ-C30, COMPASS-31, PROMIS-29, PROMIS-Cog, Perceived Stress Scale
Patient-reported outcomes | Week 6
  5 questionnaires: EORTC QLQ-C30, COMPASS-31, PROMIS-29, PROMIS-Cog, Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life University; Yoram Gidron, PhD, Principal Investigator — University of Haifa
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No